CLINICAL TRIAL: NCT06375850
Title: Effects of Topical Sesame Oil in the Prevention of Chemotherapy-associated Peripheral Venous Catheter Phlebitis: Clinical Trial.
Brief Title: Effects of Topical Sesame Oil in the Prevention of Peripheral Venous Catheter Phlebitis: Clinical Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Virginia Meneses Campos, Principal Investigator, Hospital Universitario Marqués de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Effects of topical sesame oil
Record Dates: First submitted 2024-02-29; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Phlebitis
Keywords: Neoplasms; Antineoplastic Agents; Phlebitis; Sesame Oil; Catheterization; Peripheral
MeSH Terms: conditions — Phlebitis; Neoplasms | interventions — Sesame Oil; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will be administered 2 drops of sesame oil daily along the channeled vein, about 3 centimeters from the insertion point.
  Interventions: Other: Sesame oil
- Control (Placebo Comparator): This arm will be administered 2 drops of physiological saline daily along the channeled vein, about 3 centimeters from the insertion point.
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Sesame oil — A peripheral venous catheter will be channeled to the patient admitted to the unit and who requires it. The indications included in the guide for channeling venous access of the Marqués de Valdecilla hospital will be followed.
  Once the venous access has been channeled, it will be fixed with, leaving the puncture point visible for future monitoring.
  The sesame oil chosen for the project is "Sesame bio - 100% pure vegetable oil from the Naissance brand.
  To perform the procedure, two drops of sesame oil will be applied daily by the nurse in charge of the patient during the morning shift in the area about 2 cm above the insertion point and coinciding with the course of the vein channeled for intravenous therapy. A small massage of the area of application will be performed, with an approximate extension of 3x3cm, until its absorption. It will be left to dry in the air.
  Arms: Intervention
Other: Saline solution — After cannulation of the vein following the same procedure as explained in the intervention arm, patients belonging to the control arm will be administered two drops of saline solution.
  Arms: Control

SUMMARY:
Cancer is a disease that, despite having a higher cure rate, is currently on the rise, with an increase in the number of diagnoses.

For the treatment of these patients a venous access is required, which in the first treatments is of peripheral insertion. These peripheral venous catheter in combination with the highly aggressive treatments for the veins are the cause of the appearance of chemical phlebitis.

Phlebitis is an inflammation caused by a combination of factors, whether chemical, perfusion of irritating medication; mechanical, due to the puncture site, type and fixation of the catheter and infectious, caused by the colonization of pathogenic agents whose origin is the skin and that migrate inward.

Phlebitis involves an injury to the wall of the vein, and consequently, the patient will also be at risk of thrombus formation, which in turn leads to thrombophlebitis, deep vein thrombosis or pulmonary embolism.

The existence of phlebitis involves intense and constant pain, with increased sensitivity and a sensation of heat and swelling.

With the use of topical sesame oil, and thanks to its anti-inflammatory properties, the investigators intend to study whether it is effective in preventing the appearance of phlebitis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age.
* To be conscious and have a cognitive state that allows him/her to give consent to participate in the study.
* Be diagnosed with a neoplasm that requires chemotherapy treatment.
* To be a carrier of a CVP in the upper extremity as vascular access for chemotherapy administration.

Exclusion Criteria:

* Being allergic to sesame oil.
* Be allergic to nuts.
* Not being able to speak, read and write in Spanish.
* Last days or palliative situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2025-02-11 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Number of phlebitis in oncology patients with peripheral catheter to whom sesame oil is applied topically | one year
  Sesame oil will be applied in the intervention groups, with the aim of assessing whether its application decreases the occurrence of phlebitis in oncology patients with irritating and high osmolarity intravenous medication.

SECONDARY OUTCOMES:
Other adverse effects that appear in relation to the topical application of sesame oil in patients with peripheral catheters | one year
  Registration of other adverse effects related to chemotherapy administration through a peripheral catheter: extravasation, number of cannulations during admission, catheter duration and reason for withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Meneses Campos, Principal Investigator — Employee; Virginia Meneses, Study Director — Employee
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

REFERENCES:
- [Background] Urbanetto Jde S, Peixoto CG, May TA. Incidence of phlebitis associated with the use of peripheral IV catheter and following catheter removal. Rev Lat Am Enfermagem. 2016 Aug 8;24:e2746. doi: 10.1590/1518-8345.0604.2746. PMID 27508916
- [Background] Wu XF, Yu YJ, Ying LM, Tan WF, Zhan XY, Wang LC. Hot Compress with Chinese Herbal Salt Packets Reducing PICC Catheter Complications: A Randomized Controlled Trial. Chin J Integr Med. 2018 Nov;24(11):809-814. doi: 10.1007/s11655-018-2913-y. Epub 2018 Jun 27. PMID 29946873
- [Background] Saini V, Samra T, Ahuja N, Sethi S. A prospective randomized study to evaluate safety and efficacy of heparin topical solution (1000 IU/ml) compared to heparin topical gel (200 IU/g) in prevention of infusion-associated phlebitis. Indian J Pharmacol. 2018 Nov-Dec;50(6):344-349. doi: 10.4103/ijp.IJP_201_17. PMID 30783328
- [Background] Behnamfar N, Parsa Yekta Z, Mojab F, Kazem Naeini SM. The effect of nigella sativa oil on the prevention of phlebitis induced by chemotherapy: a clinical trial. Biomedicine (Taipei). 2019 Sep;9(3):20. doi: 10.1051/bmdcn/2019090320. Epub 2019 Aug 27. PMID 31453801
- [Background] Bagheri-Nesami M, Shorofi SA, Hashemi-Karoie SZ, Khalilian A. The effects of sesame oil on the prevention of amiodarone-induced phlebitis. Iran J Nurs Midwifery Res. 2015 May-Jun;20(3):365-70. PMID 26120338
- [Background] Bigdeli Shamloo MB, Nasiri M, Maneiy M, Dorchin M, Mojab F, Bahrami H, Naseri MS, Kiarsi M. Effects of topical sesame (Sesamum indicum) oil on the pain severity of chemotherapy-induced phlebitis in patients with colorectal cancer: A randomized controlled trial. Complement Ther Clin Pract. 2019 May;35:78-85. doi: 10.1016/j.ctcp.2019.01.016. Epub 2019 Feb 2. PMID 31003690
- [Background] Goulart CB, Custodio CS, Vasques CI, Ferreira EB, Diniz Dos Reis PE. Effectiveness of topical interventions to prevent or treat intravenous therapy-related phlebitis: A systematic review. J Clin Nurs. 2020 Jul;29(13-14):2138-2149. doi: 10.1111/jocn.15266. Epub 2020 May 20. PMID 32324314
- [Background] Nekuzad N, Ashke Torab T, Mojab F, Alavi-Majd H, Azadeh P, Ehtejab G. Effect of external use of sesame oil in the prevention of chemotherapy-induced phlebitis. Iran J Pharm Res. 2012 Fall;11(4):1065-71. PMID 24250538
- [Background] Liu B, Wu Z, Lin C, Li L, Kuang X. Applicability of TIVAP versus PICC in non-hematological malignancies patients: A meta-analysis and systematic review. PLoS One. 2021 Aug 3;16(8):e0255473. doi: 10.1371/journal.pone.0255473. eCollection 2021. PMID 34343193
- See also: National Cancer Institute — https://www.cancer.gov/
- See also: Spanish Society of Medical Oncology — https://seom.org/